CLINICAL TRIAL: NCT04199754
Title: Pilot Study of Intravenous Contrast-Enhanced Cone Beam Computed Tomography (CT) in Patients Receiving Radiotherapy
Brief Title: IV Contrast-Enhanced Cone Beam Computed Tomography (CBCT) in Radiotherapy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow accrual rate due to national contrast shortage
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, David P. Horowitz, M.D., Assistant Professor of Radiation Oncology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAS0632
Record Dates: First submitted 2019-12-05; First posted 2019-12-16 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Pelvic Cancer; Abdominal Cancer
Keywords: CBCT- Cone Beam CT
MeSH Terms: conditions — Pelvic Neoplasms | interventions — Iohexol; Solutions; Injections; Radiotherapy; Saline Solution

STUDY DESIGN:
Intervention Model Description: Subjects will receive contrast enhanced CBCT prior to RT treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Contrast Enhanced Cone Beam CT (Experimental): 60 seconds after the start of the administration of IV contrast, cone beam CT will be initiated.
  Interventions: Drug: Omnipaque 300mg/mL Solution for Injection; Radiation: Cone Beam CT; Radiation: Radiation Therapy; Drug: 0.9% Saline

INTERVENTIONS:
Drug: Omnipaque 300mg/mL Solution for Injection — Prior to the contrast enhanced Cone Beam CT, 100mL of Omnipaque will be administered by IV at a rate of 2mL per second, followed by administration of 50mL of 0.9% saline.
  Other Names: Iohexol
Radiation: Cone Beam CT — 60 seconds after contrast administration, a Cone Beam CT will be performed.
Radiation: Radiation Therapy — Standard of Care Radiation Therapy will be administered, dosage depends on the type of tumor being treated.
Drug: 0.9% Saline — 50 ML of 0.9% Saline will be administered immediately after Omnipaque administration
  Other Names: Saline Solution

SUMMARY:
The purpose of this study is to find out if giving intravenous (IV) contrast (a liquid that helps with the visibility of organs and blood vessels that is given through the vein with the use of a hollow needle) during a Cone Beam Computed Tomography (CBCT- a type of computerized X-ray) can help people who have image guided radiation therapy (IGRT) for the treatment of abdominal and pelvic tumors.

DETAILED DESCRIPTION:
The goal of this pilot study is to determine the feasibility and utility of administering IV contrast during a Cone Beam Computed Tomography (CBCT) in subjects who have image guided radiation therapy (IGRT) for the treatment of abdominal and pelvic tumors. Participant duration is one visit.

Subjects will be required to fast for at least 2 hours prior to study procedures, as determined by the treating physician based on the site to be irradiated. An 18- to 22-gauge peripheral IV will be placed in the subject's arm prior to being brought to clinical treatment room. The patient will be placed in position for radiotherapy as per standard of care and will be connected to IV contrast injector. Standard of care IGRT techniques will be performed to confirm correct positioning. Iodinated IV contrast will be administered and the contrast enhance cone beam CT will be initiated. Treatment will then be administered with the patient in the position determined by non-contrast cone beam CT, as per standard of care. Immediately after completion of treatment of the subject, the study physician will complete physician survey of attitude about the utility of contrast-enhanced cone beam CT.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be greater than or equal to 18 years of age.
2. Subject must be able and willing to sign a written informed consent document.
3. Subject requiring image-guided external beam radiotherapy to abdominal or pelvic tumor with cone beam CT deemed clinically necessary by the treating physician.
4. No history of prior allergic reaction to intravenous CT contrast medium.
5. Creatinine of less than 1.9 mg/dL measured within one month prior to enrollment on the study.
6. No administration of intravenous contrast within 24 hours of administration of intravenous contrast on protocol.
7. Ability to complete New York Presbyterian Hospital iodinated contrast media administration questionnaire.
8. Negative pregnancy test for females of childbearing potential, in accordance to institutional guidelines.
9. Ability to fast for at least 2 hours prior to study procedures.
10. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-3.

Exclusion Criteria:

1. Known allergy to iohexol or any iodinated intravenous contrast medium.
2. Fluid overload that would contraindicate bolus administration of intravenous contrast.
3. Pregnant or nursing subjects.
4. Presence of single kidney or transplanted kidney
5. Acute renal failure
6. Chronic renal insufficiency, stage IV or V.
7. Administration of iodinated intravenous CT contrast medium within 24 hours of study procedures.
8. Inability to fast for at least 2 hours prior to study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Physician Survey of attitude about the utility of contrast-enhanced cone beam CT | Up to 18 Months
  The Radiation Oncologist treating physician will complete a physician survey using a Likert scale regarding attitude about the utility of contrast enhanced cone beam CT.
Blinded Match between contrast and non-contrast enhanced CBCT | Up to 18 Months
  After completion of study procedures of all enrolled subjects, images from both contrast-enhanced and non-contrast cone beam CT will undergo blinded matching by two additional study physicians. The magnitude of proposed shifts (measured in millimeters in x-, y- and z- axes) for each cone beam CT will be recorded and interrater reliability will be assessed for concordance.

CONTACTS AND LOCATIONS:
Overall Officials: David Horowitz, MD, Principal Investigator — Assistant Professor of Radiation Oncology at Columbia University Medical Center
Locations (1):
- Columbia University Irving Medical Center/Department of Radiation Oncology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katz MHG, Ou FS, Herman JM, Ahmad SA, Wolpin B, Marsh R, Behr S, Shi Q, Chuong M, Schwartz LH, Frankel W, Collisson E, Koay EJ, Hubbard JM, Leenstra JL, Meyerhardt J, O'Reilly E; Alliance for Clinical Trials on Oncology. Alliance for clinical trials in oncology (ALLIANCE) trial A021501: preoperative extended chemotherapy vs. chemotherapy plus hypofractionated radiation therapy for borderline resectable adenocarcinoma of the head of the pancreas. BMC Cancer. 2017 Jul 27;17(1):505. doi: 10.1186/s12885-017-3441-z. PMID 28750659
- [Background] Murphy JD, Adusumilli S, Griffith KA, Ray ME, Zalupski MM, Lawrence TS, Ben-Josef E. Full-dose gemcitabine and concurrent radiotherapy for unresectable pancreatic cancer. Int J Radiat Oncol Biol Phys. 2007 Jul 1;68(3):801-8. doi: 10.1016/j.ijrobp.2006.12.053. Epub 2007 Mar 26. PMID 17379445
- [Background] Krishnan S, Chadha AS, Suh Y, Chen HC, Rao A, Das P, Minsky BD, Mahmood U, Delclos ME, Sawakuchi GO, Beddar S, Katz MH, Fleming JB, Javle MM, Varadhachary GR, Wolff RA, Crane CH. Focal Radiation Therapy Dose Escalation Improves Overall Survival in Locally Advanced Pancreatic Cancer Patients Receiving Induction Chemotherapy and Consolidative Chemoradiation. Int J Radiat Oncol Biol Phys. 2016 Mar 15;94(4):755-65. doi: 10.1016/j.ijrobp.2015.12.003. Epub 2015 Dec 11. PMID 26972648
- [Background] Crane CH. Hypofractionated ablative radiotherapy for locally advanced pancreatic cancer. J Radiat Res. 2016 Aug;57 Suppl 1(Suppl 1):i53-i57. doi: 10.1093/jrr/rrw016. Epub 2016 Mar 29. PMID 27029741
- [Background] Jones B, Altunbas C, Kavanagh B, Miften M. WE-G-217BCD-08: Image Quality Effects of Dynamic Iodine Concentrations for Contrast-Enhanced Cone-Beam CT. Med Phys. 2012 Jun;39(6Part28):3974. doi: 10.1118/1.4736216. PMID 28519608
- [Background] Klostranec JM, Ehtiati T, Rao S, Radvany MG. Comparison of aortic arch and intravenous contrast injection techniques for C-arm cone beam CT: implications for cerebral perfusion imaging in the angiography suite. Acad Radiol. 2013 Apr;20(4):509-18. doi: 10.1016/j.acra.2012.10.008. PMID 23498995
- [Background] Eccles CL, Tse RV, Hawkins MA, Lee MT, Moseley DJ, Dawson LA. Intravenous contrast-enhanced cone beam computed tomography (IVCBCT) of intrahepatic tumors and vessels. Adv Radiat Oncol. 2016 Jan 26;1(1):43-50. doi: 10.1016/j.adro.2016.01.001. eCollection 2016 Jan-Mar. PMID 28740872